CLINICAL TRIAL: NCT00594087
Title: Eszopiclone for Improving Sleep Continuity in MS Patients With Sleep Disturbances and Its Impact on Daytime Fatigue
Brief Title: Eszopiclone for Improving Sleep in Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Hrayr Attarian MD Principal investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHRMS 05-255; Sepracor Study ESRC016
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2008-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Sleep Initiation and Maintenance Disorders; Fatigue
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Lunesta 2 or 3 mg
  Interventions: Drug: eszopiclone
- 2 (Placebo Comparator): Placebo 2mg or 3 mg
  Interventions: Other: placebo

INTERVENTIONS:
Drug: eszopiclone — eszopiclone 2mg or 3mg at bedtime
  Other Names: Lunesta
  Arms: 1
Other: placebo — 2 mg or 3 mg at bedtime
  Arms: 2

SUMMARY:
The purpose of this study is to determine if people with multiple sclerosis (MS) and fatigue have disrupted sleep, as was suggested in previous studies, and whether treating the disruptions of sleep improves the fatigue.

Eszoplicone, a new drug FDA approved for the treatment of insomnia, will be used to control sleep disturbances in MS patients with fatigue.

The study will last 7 weeks, 5 of which will involve being on medication. You will take eszopiclone or placebo (sugar pill), keep a sleep diary and wear an actigraph, a device about the size of a digital watch that monitors and records sleep activity. You will randomly be chosen to get either placebo or medication. Half the subjects will get placebo and half eszopiclone. The decision will be made by a pharmacist (who does not know you) according to a randomization table. Neither you nor the investigating physician will know whether you are on sugar pill or medication. At both the beginning and the conclusion of the study you will be asked to fill out 2 questionnaires to evaluate fatigue and depression and undergo some memory and speech tests. The testing will take about 2 hours. Actigraphy is a wrist-worn, watch like device that records activity during waking and sleeping without application of any sensors. It consists of a movement detector, so it can record movement and non-movement data for a week or two. You should wear it continuously during wakefulness and sleep as you go about routine daily activities. You should only take it off if you are going to shower, bathe or swim. A sleep log is a graph on which, for 2 to 3 weeks, you will record bedtime, approximate sleep time, times and duration of awakenings during the sleep period, final awakening time, and naps taken during the day to the best of your knowledge. You will also be asked to avoid getting pregnant. If you are a woman who may have the potential to get pregnant then a pregnancy test may be performed at the beginning of the study, before you receive the medication, at the first follow up visit and when you end the study.

DETAILED DESCRIPTION:
The purpose of this study is to determine if people with multiple sclerosis (MS) and fatigue have disrupted sleep, as was suggested in previous studies, and whether treating the disruptions of sleep improves the fatigue.

Eszoplicone, a new drug FDA approved for the treatment of insomnia, will be used to control sleep disturbances in MS patients with fatigue.

The study will last 7 weeks, 5 of which will involve being on medication. You will take eszopiclone or placebo (sugar pill), keep a sleep diary and wear an actigraph, a device about the size of a digital watch that monitors and records sleep activity. You will randomly be chosen to get either placebo or medication. Half the subjects will get placebo and half eszopiclone. The decision will be made by a pharmacist (who does not know you) according to a randomization table. Neither you nor the investigating physician will know whether you are on sugar pill or medication. At both the beginning and the conclusion of the study you will be asked to fill out 2 questionnaires to evaluate fatigue and depression and undergo some memory and speech tests. The testing will take about 2 hours. Actigraphy is a wrist-worn, watch like device that records activity during waking and sleeping without application of any sensors. It consists of a movement detector, so it can record movement and non-movement data for a week or two. You should wear it continuously during wakefulness and sleep as you go about routine daily activities. You should only take it off if you are going to shower, bathe or swim. A sleep log is a graph on which, for 2 to 3 weeks, you will record bedtime, approximate sleep time, times and duration of awakenings during the sleep period, final awakening time, and naps taken during the day to the best of your knowledge. You will also be asked to avoid getting pregnant. If you are a woman who may have the potential to get pregnant then a pregnancy test may be performed at the beginning of the study, before you receive the medication, at the first follow up visit and when you end the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ages 18 - 64 inclusive.
2. Female subjects must be surgically sterile, at least 1 year post menopausal, or agree to use a medically acceptable form of birth control throughout the study and for 2 weeks following the last study visit.
3. Diagnosis of relapsing-remitting MS
4. MS and MS symptoms must be stable (no evidence of worsening or of exacerbations) for at least 3 months prior to screening visit. The date of last recorded exacerbation will be captured at enrollment.
5. EDSS score </= 5
6. Diagnosis of fatigue based on fatigue questionnaires, specifically the Fatigue Descriptive Scale (FDS) in which a score of five higher is considered to be indicative of fatigue (range 0-13)
7. Actigraphic evidence of sleep disturbances defined a sleep latency of 30 minutes or longer, and/or total sleep time of less than 6.5 hours.
8. Finally a CESD score of under 20 (20 or more is suggestive of Major Depression)

Exclusion Criteria:

1. Pregnant and breast-feeding women
2. Subjects with any history of substance and/or alcohol abuse or dependence within 5 years prior to screening.
3. Subjects who are the sole caretaker of infants and young children because they may be too sedated in the middle of the night in case they need to get up and take care of an infant or a child.
4. Patients with past history of allergy to eszopiclone or Zopiclone.
5. Patients with primary progressive Multiple Sclerosis.
6. Subjects with impaired cognition as measured by Mini Mental State Examination (MMSE) score of 26 or less
7. Subjects with history suggestive of another primary sleep disorder including OSAS, PLMS, or RLS
8. Any patients with any known active DSM-IV axis I (i.e. schizophrenia, etc) or any other psychiatric disorder which would compromise the investigator's ability to evaluate the safety and efficacy of the study medication.
9. Patients 65 years old and older because the drug at the 3 mg dose has not been FDA approved to be used in this age group.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Fatigue | 7 weeks

SECONDARY OUTCOMES:
Sleep continuity | 7 weeks
Neurocognitive function | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hrayr Attarian, MD, Principal Investigator — UVM
Locations (1):
- University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Background] Attarian HP, Brown KM, Duntley SP, Carter JD, Cross AH. The relationship of sleep disturbances and fatigue in multiple sclerosis. Arch Neurol. 2004 Apr;61(4):525-8. doi: 10.1001/archneur.61.4.525. PMID 15096400
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Background] Jean-Louis G, Mendlowicz MV, Gillin JC, Rapaport MH, Kelsoe JR, Zizi F, Landolt H, von Gizycki H. Sleep estimation from wrist activity in patients with major depression. Physiol Behav. 2000 Jul 1-15;70(1-2):49-53. doi: 10.1016/s0031-9384(00)00228-6. PMID 10978477
- [Background] Iriarte J, Katsamakis G, de Castro P. The Fatigue Descriptive Scale (FDS): a useful tool to evaluate fatigue in multiple sclerosis. Mult Scler. 1999 Feb;5(1):10-6. doi: 10.1177/135245859900500103. PMID 10096097
- See also: University of Vermont — http://www.uvm.edu